CLINICAL TRIAL: NCT01891903
Title: TO TRANSLATE AND VALIDATE THE ToPAS (TORONTO PSORIATIC SCREENING QUESTIONNAIRE) FOR THE SCREENING OF PSORIATHIC ARTHRITIS PATIENTS IN DERMATOLOGY CLINICS
Brief Title: to Translate and Validate the TOPAS TORONTO PSORIATIC SCREENING QUESTIONNAIRE)Into Spanish
Acronym: spanishTopas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Reumatologia Integral LTDA (Other)
Responsible Party: Principal Investigator, Adriana Beltran, ADRIANA BELTRAN OSTOS, Reumatologia Integral LTDA
Other Study IDs: TOPAS52424166
Record Dates: First submitted 2013-06-18; First posted 2013-07-03 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-06

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Days
Oversight: Data Monitoring Committee: Yes

SUMMARY:
TO TRANSALETE AND VALIDATE DE TORONTO PSORIATIC ARTHRITIS SECREENING QUESTIONAIRE INTO SPANISH

DETAILED DESCRIPTION:
THIS IS PART OF THE COLOMBIAN REGISTRY OF PATIENTS WITH PSORIASIS AND PSORIATIC ARTHRITIS

ELIGIBILITY:
Inclusion Criteria:

* ADULT WITH PSORIASIS IN THE DERMATOLOGY CLINIC

Exclusion Criteria:

* ADULT WITH OTHER AUTOIMMUNE DISEASE

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PATIENTS WITH PSORIASIS ASESSED IN THE DERMATOLOGY CLINIC
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-08 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
The Kuder Richardson Coefficient of reliability (K-R 20) | 4 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fernandez, rheumatolo, Study Director — hospital san ignasio
Locations (1):
- Hospital Universitario Clinica San Rafael, Bogota, Cundinamarca, Colombia